CLINICAL TRIAL: NCT03671694
Title: Laser Vaginal Treatment for Stress Urinary Incontinence
Brief Title: Laser Vaginal Treatment for SUI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Sunnybrook_womens
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2023-04

CONDITIONS: Stress Urinary Incontinence
Keywords: laser treatment
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: only the care provider (who is not involved with recruitment or evaluation of patients' outcomes) will be aware of the treatment assignments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laser treatment (Active Comparator): Erbium-YAG laser treatment to the vagina
  Interventions: Procedure: Erbium-YAG laser vaginal treatment
- sham treatment (Placebo Comparator): sham treatment with laser placebo
  Interventions: Procedure: Erbium-YAG laser vaginal treatment

INTERVENTIONS:
Procedure: Erbium-YAG laser vaginal treatment — Erbium-YAG laser vaginal treatment

SUMMARY:
RCT designed to answer the question:

Does the application of Erbium: YAG laser treatment to the vagina improve urine control for women with SUI?

DETAILED DESCRIPTION:
This is a double blinded randomized controlled clinical trial with a treatment arm and a sham treatment arm followed by an open label trial at 6 months for any sham treatment arm participants who do not meet treatment success.

The primary goal is to compare the subjective success rates for the resolution of UI for the vaginal laser treatment at 6 months. Secondary aims include an assessment of complications, resolution of SUI symptoms (objective and subjective measures), patient bother from UI, quality of life and patient satisfaction. The proposed sample size is 182 patients. At the 6-month post treatment evaluation, the treatment allocation will be unmasked. The trial will be of approximately 3 years in duration (1 year to recruit and 2 years for follow up).

ELIGIBILITY:
Inclusion Criteria:

1. Female patient, aged 18 years or older at the time of enrollment,
2. primary symptoms of SUI, as confirmed by patient medical history and clinical symptoms, including a focused incontinence evaluation; for a duration of at least 3 months (patient can be rescreened after this time interval has passed).
3. The patient agrees to no new parallel treatment for SUI during the treatment period and the 6 months following it.
4. objective proof of SUI: Observation of urine leakage by cough and valsalva (positive stress test) at a bladder volume of ≤ 300cc
5. Bladder capacity ≥200cc
6. Post void residual ≤100cc with Stage I or lower pelvic organ prolapse

Exclusion Criteria:

1. Patient is pregnant, lactating, or plans to become pregnant during the course of the Study; or Patient is <12 months post partum
2. Patient has other predominant type of UI (eg Urgency UI, overflow UI, fistula)
3. Patient has a vaginal condition that does not allow proper vaginal placement of the laser probe in its protective speculum
4. Current chemo/ radiotherapy; history of pelvic radiation
5. Systemic diseases known to affect bladder function (eg Parkinson's disease, multiple sclerosis, spina bifida, spinal cord injury)
6. Current or history of urethral diverticulum, prior augmentation cystoplasty, implanted nerve stimulators for bladder symptoms
7. History of synthetic sling
8. Pelvic surgery < 3 months
9. Current evaluation or treatment for chronic pelvic pain
10. Patient has pelvic organ/ vaginal prolapse extending to or out of the vaginal opening
11. Participation in another treatment intervention that might interfere with the results of this trial
12. Patient has a medical condition or disorder that may limit life expectancy or that may cause non-compliance with the protocol (e.g. unable to perform self-evaluations and/or accurately report medical history, urinary symptoms, and/or data).
13. Patient has ambulatory 24 hour pad test, where the increased pad weight is < 3 grams.
14. Patient is non-ambulatory (ambulatory with assistive devices allowed)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
SUI cure | 6 months post treatment
  ICIQ questionnaire: The International Consultation on Incontinence Questionnaire (ICIQ) is a subjective measure of the severity of urinary loss and quality of life for those with incontinence.
  With the short form, there are 3 questions with a multi-choice selection of responses with each response having an assigned score. The total score (additive from the 3 questions) are between 0 - 21. Higher scores are indicative of greater severity.

SECONDARY OUTCOMES:
Adverse effects | 6,12 24 months post treatment
  Number of participants with any reported adverse effects: local burn, bleeding, irritation, infection, vaginal discharge etc.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Lee, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ippolito GM, Crescenze IM, Sitto H, Palanjian RR, Raza D, Barboglio Romo P, Wallace SA, Orozco Leal G, Clemens JQ, Dahm P, Gupta P. Vaginal lasers for treating stress urinary incontinence in women. Cochrane Database Syst Rev. 2025 Jul 25;7(7):CD013643. doi: 10.1002/14651858.CD013643.pub2. PMID 40709601